CLINICAL TRIAL: NCT05805943
Title: Phase I/II Study of IMM0306 in Patients With Relapsed or Refractory CD20-positive B-cell Non-Hodgkin's Lymphoma
Brief Title: Study of IMM0306 in Patients With Relapsed or Refractory CD20-positive B-cell Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM0306-I
Record Dates: First submitted 2023-03-24; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: CD20-positive B-cell Non-Hodgkin's Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMM0306 Monotherapy (Experimental): Phase I dose escalation part, participants with relapsed or refractory CD20-positive B-cell non-Hodgkin's lymphoma (B-NHL) will be enrolled to receive IMM0306. The dose of IMM0306 will depend on when you join this study. About 1-6 participants will be enrolled at each dose level.
  Phase II dose expansion part, participants will receive IMM0306 at the recommended dose that was found in dose escalation part.
  Interventions: Drug: IMM0306

INTERVENTIONS:
Drug: IMM0306 — IMM0306 is an bi-specific antibody

SUMMARY:
This is a Phase I/II, Single-Arm, Open-Label, Multicentre Study to Evaluate the Safety and Efficacy of IMM0306 in Patients with Relapsed or Refractory B-Cell Non- Hodgkin's Lymphoma (R/R B-NHL).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CD20-positive B-cell non-Hodgkin's lymphoma (B-NHL) that has been diagnosed, including but not limited to diffuse large B-cell lymphoma (DLBCL) Follicular lymphoma (FL), mucosal lymphoma (MALT-L), small lymphocytic lymphoma (SLL) / chronic lymphocytic leukemia (CLL).
* At least one measurable or assessable tumor lesion.
* Adequate organ and hematologic function.
* Eastern Co-operative Oncology Group (ECOG) score 0 to 2.
* All adverse events from prior treatment must be CTCAE v5.0 grade <= 1

Exclusion Criteria:

* Active central nervous system (CNS) lymphoma.
* Systemic steroid therapy (dose equivalent to > 10 mg prednisone / day).
* History of severe allergic reactions to macromolecular protein preparations/monoclonal antibodies and any test drug components (CTCAE v5.0 grade >=3).
* Have evidence of severe uncontrollable active infection.
* Subjects have deep vein embolism or pulmonary embolism within 6 months before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Evaluated for DLTs during the first 28-day cycle
Complete response rate | up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang J, Song Y, Zhou K, Li Z, Zhang M, Jing H, Wang Z, Yu L, Meng W, Lu Q, Tian W, Shi Y. Safety and efficacy of amulirafusp alfa (IMM0306), a fusion protein of CD20 monoclonal antibody with the CD47 binding domain of SIRPalpha, in patients with relapsed or refractory B-cell non-Hodgkin lymphoma: a phase 1/2 study. J Hematol Oncol. 2024 Dec 18;17(1):123. doi: 10.1186/s13045-024-01646-2. PMID 39696680